CLINICAL TRIAL: NCT03004924
Title: A Phase 3, Multi-center, Randomized, Double-Masked Study to Evaluate the Clinical Efficacy and Safety of SHP640 (PVP-Iodine 0.6% and Dexamethasone 0.1%) Ophthalmic Suspension Compared to Placebo in the Treatment of Bacterial Conjunctivitis
Brief Title: Treatment of Bacterial Conjunctivitis With SHP640 Compared to PVP-Iodine and Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHP640-303; 2016-003361-25 (EudraCT Number)
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Results first posted 2019-10-28 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SHP640 (Experimental): Participants will instill 1 drop of SHP640 (povidone-iodine [PVP-I] 0.6 percent [%] and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times daily (QID) for 7 days.
  Interventions: Drug: SHP640
- PVP-I 0.6% (Active Comparator): Participants will instill 1 drop of PVP-I 0.6% ophthalmic solution in each eye 4 times QID for 7 days
  Interventions: Drug: PVP-I 0.6%
- Placebo (Placebo Comparator): Participants will instill 1 drop of placebo ophthalmic solution in each eye 4 times QID for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHP640 — Instill 1 drop of SHP640 (povidone-iodine [PVPI] 0.6% and Dexamethasone 0.1%) ophthalmic suspension in each eye QID (with a minimum of 2 hours between doses) for 7 days.
  Arms: SHP640
Drug: PVP-I 0.6% — Instill 1 drop of PVP-I 0.6% ophthalmic solution in each eye 4 times QID (with a minimum of 2 hours between doses) for 7 days.
  Arms: PVP-I 0.6%
Drug: Placebo — Instill 1 drop of placebo ophthalmic solution in each eye 4 times QID (with a minimum of 2 hours between doses) for 7 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if an investigational treatment is effective compared with placebo and PVP-Iodine in the treatment of adults and children with bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* An understanding, ability, and willingness to fully comply with study procedures and restrictions (by the parent(s), guardian, or legally authorized representative, if applicable).
* Ability to voluntarily provide written, signed, and dated (personally or via a parent(s), guardian, or legally authorized representative(s) informed consent (and assent, if applicable) to participate in the study.
* Participants of any age at Visit 1 (Note: participants less than (<) 3 months of age at Visit 1 must have been full-term, that is (ie,) greater than or equal to (>=) 37 weeks gestational age at birth).
* Have a negative AdenoPlus® test in both eyes within 24 hours of Visit 1 or at Visit 1.
* Have a clinical diagnosis of suspected bacterial conjunctivitis in at least 1 eye confirmed by the presence of the following minimal clinical signs and symptoms in that same eye:

  1. Report presence of signs and/or symptoms of bacterial conjunctivitis for less than or equal to (<=) 4 days prior to Visit 1
  2. Bulbar conjunctival injection: a grade of >= 1 on 0-4 scale of Bulbar Conjunctival Injection Scale
  3. Ocular conjunctival discharge: a grade of >= 1 (mild) on a 0-3 scale of Ocular Conjunctival Discharge Scale
* Be willing to discontinue contact lens wear for the duration of the study.
* Have a Best Corrected Visual Acuity (BCVA) of 0.60 logMAR or better in each eye as measured using an Early Treatment Diabetic Retinopathy Study (ETDRS) chart. BCVA will be assessed by an age appropriate method in accordance with the AAP Policy Statement for Visual System Assessment in Infants, Children, and Young Adults by Pediatricians (Donahue and Baker, 2016; American Academy of Pediatrics, 2016). The policy statement recommends formal vision screening can begin at 3 years of age. VA measurements for children under the age of 3 will be done at the discretion of the investigator. If not done, child should be able to fixate on and follow a moving object, except participants < 2 months of age who have not yet developed this ability. Participants < 2 months will be enrolled at the discretion of investigator.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.

Exclusion Criteria:

* Current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinical or laboratory assessments, per investigator's discretion.
* Current or relevant history of physical or psychiatric illness, any medical disorder that may make the participant unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
* Have known or suspected intolerance or hypersensitivity to the investigational product, closely related compounds, or any of the stated ingredients.
* Prior enrollment in a FST-100 or SHP640 clinical study.
* Participants who are employees, or immediate family members of employees (who are directly related to study conduct), at the investigational site.
* Have a history of ocular surgical intervention within <= 6 months prior to Visit 1 or planned for the period of the study.
* Have a preplanned overnight hospitalization during the period of the study.
* Have presence of any intraocular, corneal, or conjunctival ocular inflammation (example [eg,] uveitis, iritis, ulcerative keratitis, chronic blepharoconjunctivitis), other than bacterial conjunctivitis.
* Have active or a history of ocular herpes.
* Have at enrollment or within <= 30 days of Visit 1, a clinical presentation more consistent with the diagnosis of non-infectious conjunctivitis (except presumed seasonal/perennial allergic conjunctivitis) or non-bacterial ocular infection (eg, viral, fungal, acanthamoebal, or other parasitic). Note: history or concomitant presence of presumed seasonal or perennial allergic conjunctivitis signs/symptoms is not exclusionary.
* Neonates or infants (ie, participants less than 12 months of age) who have suspected or confirmed (based on the result of any test conducted prior to screening) conjunctivitis of gonococcal, chlamydial, herpetic or chemical origin.
* Neonates or infants (ie, participants less than 12 months of age) whose birth mothers had any sexually transmitted disease within 1 month of delivery or any history of genital herpes.
* Presence of nasolacrimal duct obstruction at Visit 1 (Day 1).
* Presence of any significant ophthalmic condition (eg, Retinopathy of Prematurity, congenital cataract, congenital glaucoma) or other congenital disorder with ophthalmic involvement that could affect study variables.
* Be a known intraocular pressure (IOP) steroid responder, have a known history or current diagnosis of glaucoma or be a glaucoma suspect.
* Have any known clinically significant optic nerve defects.
* Have a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome; presence of corneal epithelial defect or any significant corneal opacity at Visit 1.
* Presence of significant, active condition in the posterior segment that requires invasive treatment (eg, intravitreal treatment with vascular endothelial growth factor inhibitors or corticosteroids) and may progress during the study participation period.
* Have used any topical ocular or systemic antibiotics within <= 7 days of enrollment.
* Have used any topical ocular non-steroidal anti-inflammatory drugs within <= 1 day of enrollment.
* Have used any topical ophthalmic steroids in the last <= 14 days.
* Have used any systemic corticosteroid agents within <= 14 days of Day 1. Stable (initiated >= 30 days prior to enrollment) use of inhaled and nasal corticosteroids is allowed, given no anticipated change in dose for the duration of the study. Topical dermal steroids are allowed except in the periocular area.
* Have used non-corticosteroid immunosuppressive agents within <= 14 days of Day 1.
* Have used any topical ophthalmic products, including tear substitutes, and over-the-counter preparations such as lid scrubs, within 2 hours of Visit 1 and be unable to discontinue all topical ophthalmic products for the duration of the study. Use of hot or cold compresses is also not permitted during the study.
* Have any significant ocular disease (eg, Sjogren's syndrome) or any uncontrolled systemic disease or debilitating disease (eg, cardiovascular disease, hypertension, sexually transmitted diseases/infections, diabetes, or cystic fibrosis) that may affect the study parameters, per investigator's discretion.
* Any known history of immunodeficiency disorder or known active conditions predisposing to immunodeficiency, such as human immunodeficiency virus, hepatitis B or C, evidence of active hepatitis A (anti-hepatitis A virus immunoglobulin M), or organ or bone marrow transplantation.
* Within 30 days prior to the first dose of investigational product:

  1. Have used an investigational product or device, or
  2. Have been enrolled in a clinical study (including vaccine studies) that, in the investigator's opinion, may impact this Shire-sponsored study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 753 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (163):
- United States (125):
  - Arizona Eye Center, Chandler, Arizona
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - M&M Eye Institute, Prescott, Arizona
  - Schwartz Laser Eye Center, Scottsdale, Arizona
  - Walman Eye Center, Sun City, Arizona
  - Milton M. Hom, OD, FAAO, Azusa, California
  - Clark S Tsai Eye Center, Concord, California
  - Lugene Eye Institute Inc, Glendale, California
  - Mark B. Kislinger, MD, Inc., Glendora, California
  - Inland Eye Specialists, Hemet, California
  - Lakeside Vision Center, Irvine, California
  - Hull Eye Center, Lancaster, California
  - Eye Physicians of Long Beach, Long Beach, California
  - Oxford Optical, Los Angeles, California
  - Sok H. Nam, M.D. Inc., Los Angeles, California
  - University of Southern California, Los Angeles, California
  - Macy Eye Center, Los Angeles, California
  - North Valley Eye Medical Group Inc, Mission Hills, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - Arch Health Partners, Poway, California
  - Martel Eye Medical Group, Rancho Cordova, California
  - Shasta Eye Medical Group, Inc., Redding, California
  - Clinical Trials Research, Roseville, California
  - Sacramento Eye Consultants, Sacramento, California
  - WCCT Global (PH 1 Unit), Santa Ana, California
  - East West Eye Institute, Torrance, California
  - Wolstan & Goldberg Eye Associates, Torrance, California
  - Specialty Eye Care, Parker, Colorado
  - Danbury Eye Physicians and Surgeons, Danbury, Connecticut
  - Ophthalmic Consultants of Connecticut, Meriden, Connecticut
  - Windham Eye Group, Willimantic, Connecticut
  - The Eye Associates of Manatee, LLP, Bradenton, Florida
  - Bruce A. Segal, MD, PA, Delray Beach, Florida
  - South Florida Vision, Fort Lauderdale, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Inc., Largo, Florida
  - Millenium Clinical Research, Miami, Florida
  - Millennium Clinical Research, Inc., Miami, Florida
  - South Florida Research Center Inc., Miami, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Lorites Medical Group, Miami, Florida
  - Pediatric & Adult Research Center, LLC, Orlando, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Score Physician Alliance, LLC, St. Petersburg, Florida
  - East Florida Eye Institute, Stuart, Florida
  - Andrew Gardner Logan, MD / dba Logan Ophthalmic Research, LLC, Tamarac, Florida
  - Logan Ophthalmic Research, LLC, Tamarac, Florida
  - International Research Center, Tampa, Florida
  - Eye Care Centers Management, Inc., Morrow, Georgia
  - Jenkins Eye Care, Honolulu, Hawaii
  - Saltzer Medical Group, Nampa, Idaho
  - Wohl Eye Center, Bloomingdale, Illinois
  - Jackson Eye, Lake Villa, Illinois
  - Illinois Eye Center, Peoria, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Midwest Cornea Associates, LLC, Indianapolis, Indiana
  - Sabates Eye Centers, Leawood, Kansas
  - Kannarr Eye Care, Pittsburg, Kansas
  - Cincinnati Eye Institute, Edgewood, Kentucky
  - Koffler Vision Group, Lexington, Kentucky
  - Kentucky Eye Institute, Lexington, Kentucky
  - The Eye Care Institute, Louisville, Kentucky
  - Dr. Haider Eye Care, Louisville, Kentucky
  - Senior Health Services, Louisville, Kentucky
  - Baker, Carl W, Paducah, Kentucky
  - Lakeview Vision, Gretna, Louisiana
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Eye Center Northeast, Bangor, Maine
  - Massachusetts Eye and Ear Infirmary, Boston, Massachusetts
  - NECCR PrimaCare Research, Fall River, Massachusetts
  - Shire Call Center, Lexington, Massachusetts
  - Clinical Eye Research of Boston, Winchester, Massachusetts
  - Minnesota Eye Consultants, P.A, Bloomington, Minnesota
  - Lifelong Vision Foundation, Chesterfield, Missouri
  - Silverstein Eye Centers, Kansas City, Missouri
  - Moyes Eye Center, Kansas City, Missouri
  - Mercy Research, Springfield, Missouri
  - Washington University, St Louis, Missouri
  - Tekwani Vision Center, St Louis, Missouri
  - Ophthalmology Associates, St Louis, Missouri
  - Opthalmology Consultants Ltd., St Louis, Missouri
  - NV Eye Physicians, Henderson, Nevada
  - Wellish Vision Institute, Las Vegas, Nevada
  - Emil A. Stein, M.D., Ltd., Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Farkas, Kassalow, Resnick &Associates, New York, New York
  - Fichte, Endl& Elmer Eyecare, Niagara Falls, New York
  - South Shore Eye Care, Wantagh, New York
  - Oculus Research at Garner EyeCareCenter, Raleigh, North Carolina
  - James Branch, M.D., Winston-Salem, North Carolina
  - Apex Eye Kenwood, Cincinnati, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Apex Eye, Cincinnati, Ohio
  - Cleveland Eye Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Columbus Eye Center, Columbus, Ohio
  - SkyVision Centers, Westlake, Ohio
  - IPS Research Company*, Oklahoma City, Oklahoma
  - Pacific Clear Vision Institute, Eugene, Oregon
  - Matossian Eye Associates, Doylestown, Pennsylvania
  - Philadelphia Eye Associates, Philadelphia, Pennsylvania
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Wyomissing Optometric Center, Wyomissing, Pennsylvania
  - Bluestein Custom Vision, Charleston, South Carolina
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - Total Eye Care, PA, Memphis, Tennessee
  - Eye Specialty Group, Memphis, Tennessee
  - Nashville Vision Associates, Nashville, Tennessee
  - Toyos Clinic, Nashville, Tennessee
  - Eyeland Vision, El Paso, Texas
  - Houston Eye Associates, Houston, Texas
  - Advanced Laser Vision & Surgical Institute, Houston, Texas
  - Lake Travis Eye & Laser Center, Lakeway, Texas
  - DCT- Shah Research, LLC dba Discovery Clinical Trials, Mission, Texas
  - Sun Research Institute, LLC, San Antonio, Texas
  - R and R Eye Research, LLC., San Antonio, Texas
  - Lone Star Eye Care, P.A., Sugar Land, Texas
  - Ericksen Research & Development, LLC, Clinton, Utah
  - The Eye Institute of Utah, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - Chrysalis Clinical Research, St. George, Utah
  - Emerson Clinical Research Institute, Falls Church, Virginia
  - Piedmont Eye Center, Inc., Lynchburg, Virginia
  - University of Wisconsin, Madison, Wisconsin
- University of the Sunshine Coast Clinical Trials Centre, Sippy Downs, Queensland, Australia
- Austria (3):
  - Augenklinik, Studienzentrum, Kepler-Universitätsklinikum GmbH, Linz
  - AKH - Medizinische Universitaet Wien, Vienna
  - Vienna Institute for Research in Ocular Surgery, Vienna
- Canada (2):
  - The Ottawa Hospital - General Campus, University of Ottawa Eye Institute, Ottawa, Ontario
  - University of Waterloo School of Optometry and Vision Science, Waterloo, Ontario
- Estonia (3):
  - Eye Clinic Dr Kirsta Turman (Kreutzwaldi Silmakeskus), Tallinn
  - East Tallinn Central Hospital Eye Clinic, Tallinn
  - Tartu University Hospital, Tartu
- CHU Limoges - Hopital Dupuytren, Limoges, Haute Vienne, France
- Hungary (5):
  - SZTE Szemeszeti Klinika, Szeged, Csongrád megye
  - Bugat Pal Hospital Clinexpert Gyongyos, Gyöngyös, Heves County
  - Debreceni Egyetem, Debrecen
  - Kaposi Mór Hospital, Kaposvár
  - Csolnoky Ferenc Korhaz, Veszprém
- Israel (7):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Rambam MC, Haifa
  - Sharey Zedek MC, Jerusalem
  - Rabin Medical Center-Beilinson Campus., Petah Tikva
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Medical Center, Tel Aviv
- A.O.U. Policlinico San'Orsola-Malpighi, Bologna, Italy
- Poland (5):
  - Centrum Medyczne Uno-Med, Krakow, Malopolska
  - Szpital Specjalistyczny nr 1, Bytom
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - Centrum Medyczne Uno-Med, Tarnów
  - Retina Sp. z o.o., Warsaw
- Puerto Rico (3):
  - Emanuelli Research & Development Center, LLC, Arecibo
  - Centro Dotal de Investigaciones de Servicios de Salud, Carolina
  - Berrocal and Associates, San Juan
- South Africa (3):
  - Newtown Clinical Research Centre, Johannesburg, Gauteng
  - Pretoria Eye Institute, Pretoria, Gauteng
  - Into Research, Pretoria, Gauteng
- Spain (4):
  - Instituto Oftalmológico Fernández-Vega, Oviedo, Principality of Asturias
  - Clinica Oftalmologia Gil Piña, Huelva
  - Clinica Rementeria, Madrid
  - Cartujavision, Seville

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 121 centers in 14 countries between 29 Mar 2017 (first participant first visit) and 01 Oct 2018 (last participant last visit).
Pre-assignment Details: A total of 1080 participants were screened, of them 753 enrolled and randomized to treatment. One participant was randomized in error and therefore captured only in the intent-to-treat (ITT) population.
Groups:
- SHP640: Participants administered 1 drop of SHP640 (povidone-iodine [PVP-I] 0.6 percent [%] and Dexamethasone 0.1%) ophthalmic suspension in each eye 4 times a day (QID) for 7 days.
- PVP-I 0.6%: Participants administered 1 drop of PVP-I 0.6% ophthalmic solution in each eye QID for 7 days.
- Placebo: Participants administered 1 drop of placebo ophthalmic solution in each eye QID for 7 days.
Period: Overall Study
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Started | 324 | 108 | 321
Completed | 297 | 94 | 293
Not Completed | 27 | 14 | 28
Not completed — Adverse Event | 6 | 5 | 10
Not completed — Protocol Violation | 4 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 5
Not completed — Lost to Follow-up | 6 | 1 | 4
Not completed — Lack of Efficacy | 2 | 4 | 2
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Withdrawal by parent/guardian | 1 | 0 | 2
Not completed — Screen Failure | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0
Not completed — Terminated by Sponsor | 0 | 0 | 1
Not completed — Missed Study Visit | 0 | 0 | 2
Not completed — HSV1 Positive | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: ITT population included all randomized participants.
Groups:
- SHP640: Participants administered 1 drop of SHP640 ophthalmic suspension in each eye QID for 7 days.
- Total: Total of all reporting groups
Arm/Group | SHP640 | PVP-I 0.6% | Placebo | Total
Number analyzed (Participants) | 324 | 108 | 321 | 753
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.2 (22.87) | 43.1 (23.03) | 44.7 (23.00) | 44.3 (22.92)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 191 | 71 | 199 | 461
  Male | 133 | 37 | 122 | 292
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 62 | 30 | 87 | 179
  Ethnicity: Not Hispanic or Latino | 254 | 76 | 230 | 560
  Ethnicity: Not reported | 4 | 2 | 2 | 8
  Ethnicity: Other | 4 | 0 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 1 | 3 | 4
  Race: Asian | 12 | 0 | 8 | 20
  Race: Black or African American | 54 | 18 | 54 | 126
  Race: White | 250 | 88 | 250 | 588
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 2 | 2
  Race: Other | 6 | 1 | 4 | 11
  Race: Multiple | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Resolution Among Who Received SHP640 or Placebo on Day 5
Description: Clinical resolution was defined as absence (score=0) of bulbar conjunctival injection and ocular conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from validated bulbar redness (VBR) scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale. The study eye was defined as an eye with score of at least 1 for both ocular conjunctival discharge and bulbar conjunctival redness at baseline. Data analysis was performed in SHP640 and placebo reporting groups only but not in PVP-I 0.6%.
Time Frame: Day 5
Population: Modified intent-to-treat (mITT) population included participants who received at least one dose of investigational product (IP) and had a positive bacterial culture (presence of one or more bacterial species at or above pathological threshold) at baseline in the study. Analysis was done in SHP640 and placebo reporting groups only.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 220 | 0 | 222
Participants | 111 | 0 | 95
Statistical Analysis 1: Comparison: SHP640 vs Placebo; Test type: Superiority; p = 0.127, Fisher Exact; Difference in response rate = 7.7, 95% CI 2-sided [-1.6 to 16.9]

2. Secondary Outcome: Number of Participants With Bacterial Eradication Among Who Received SHP640 or Placebo on Day 5
Description: Bacterial eradication was defined as absence of all bacterial species present at or above pathological threshold at baseline in the study eye. Bacterial species were identified by Matrix Assisted Laser Desorption/Ionization-Time of Flight Mass Spectrometry, using their unique protein patterns. Pathological threshold for individual bacterial species was based on colony-forming unit (CFU)/mL threshold levels established by Cagle and modified by Leibowitz for different ocular bacterial species found in the specimens collected from each participant. Data analysis was performed in SHP640 and placebo reporting groups only but not in PVP-I 0.6%.
Time Frame: Baseline, Day 5
Population: mITT population included participants who received at least one dose of IP and had a positive bacterial culture (presence of one or more bacterial species at or above pathological threshold) at baseline in the study. Here, the number of participants analyzed refer to the participants evaluable for this outcome at specified time point.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 217 | 0 | 218
Participants | 94 | 0 | 102
Statistical Analysis 1: Comparison: SHP640 vs Placebo; Test type: Superiority; p = 0.500, Fisher Exact; Difference in response rate = -3.5, 95% CI 2-sided [-12.8 to 5.9]

3. Secondary Outcome: Number of Participants With Clinical Resolution
Description: Clinical resolution was defined as absence (score=0) of bulbar conjunctival injection and ocular conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale. The study eye was defined as an eye with score of atleast 1 for both ocular conjunctival discharge and bulbar conjunctival redness at baseline.
Time Frame: Day 3, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Participants
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | 39 | 6 | 39
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 148 | 39 | 133
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | 150 | 47 | 154

4. Secondary Outcome: Number of Participants With Bacterial Eradication
Description: Bacterial eradication was defined as absence of all bacterial species present at or above pathological threshold at baseline in the study eye. Bacterial species were identified by Matrix Assisted Laser Desorption/Ionization-Time of Flight Mass Spectrometry, using their unique protein patterns. Pathological threshold for individual bacterial species was based on CFU/mL threshold levels established by Cagle and modified by Leibowitz for different ocular bacterial species found in the specimens collected from each participant.
Time Frame: Day 3, 8 and 12
Population: mITT population included participants who received at least one dose of IP and had a positive bacterial culture (presence of one or more bacterial species at or above pathological threshold) at baseline in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Participants
  Day 3: number analyzed (Participants) | 213 | 75 | 214
  Day 3 | 76 | 33 | 79
  Day 8: number analyzed (Participants) | 205 | 64 | 200
  Day 8 | 85 | 25 | 87
  Day 12: number analyzed (Participants) | 194 | 60 | 183
  Day 12 | 83 | 21 | 82

5. Secondary Outcome: Bulbar Conjunctival Injection Score
Description: Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale.
Time Frame: Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 216 | 76 | 218
  Day 3 | 1.0 (0.84) | 1.3 (0.90) | 1.1 (0.86)
  Day 5: number analyzed (Participants) | 207 | 65 | 209
  Day 5 | 0.5 (0.77) | 0.7 (0.88) | 0.7 (0.80)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 0.3 (0.64) | 0.4 (0.61) | 0.4 (0.61)
  Day 12: number analyzed (Participants) | 196 | 62 | 187
  Day 12 | 0.2 (0.56) | 0.2 (0.47) | 0.2 (0.48)

6. Secondary Outcome: Change From Baseline in the Bulbar Conjunctival Injection Score
Description: as for outcome 5
Time Frame: Baseline, Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 216 | 76 | 218
  Day 3 | -1.0 (0.77) | -0.8 (0.76) | -0.9 (0.76)
  Day 5: number analyzed (Participants) | 207 | 65 | 209
  Day 5 | -1.5 (0.87) | -1.3 (0.99) | -1.3 (0.85)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | -1.8 (0.91) | -1.6 (0.86) | -1.6 (0.81)
  Day 12: number analyzed (Participants) | 196 | 62 | 187
  Day 12 | -1.8 (0.89) | -1.8 (0.74) | -1.8 (0.82)

7. Secondary Outcome: Ocular Conjunctival Discharge Score
Description: Ocular conjunctival discharge was assessed based on a 0 (No evidence of discharge in the conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale.
Time Frame: Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | 0.7 (0.73) | 0.8 (0.74) | 0.7 (0.76)
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | 0.3 (0.57) | 0.2 (0.44) | 0.4 (0.60)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 0.1 (0.43) | 0.1 (0.31) | 0.2 (0.47)
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | 0.1 (0.49) | 0.0 (0.22) | 0.1 (0.28)

8. Secondary Outcome: Change From Baseline in the Ocular Conjunctival Discharge Score
Description: as for outcome 7
Time Frame: Baseline, Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | -0.9 (0.77) | -0.8 (0.67) | -0.9 (0.85)
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | -1.4 (0.74) | -1.4 (0.75) | -1.3 (0.75)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | -1.5 (0.71) | -1.5 (0.73) | -1.4 (0.74)
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | -1.5 (0.76) | -1.6 (0.71) | -1.6 (0.73)

9. Secondary Outcome: Global Clinical Score
Description: Global clinical score was defined as the sum of bulbar conjunctival injection and ocular conjunctival discharge scores. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale. The study eye was defined as an eye with a score of at least 1 for both ocular conjunctival discharge and bulbar conjunctival redness at baseline.
Time Frame: Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | 1.7 (1.37) | 2.1 (1.39) | 1.9 (1.42)
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | 0.8 (1.18) | 0.9 (1.19) | 1.0 (1.18)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 0.4 (0.93) | 0.5 (0.77) | 0.6 (0.93)
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | 0.4 (0.90) | 0.3 (0.55) | 0.3 (0.67)

10. Secondary Outcome: Change From Baseline in the Global Clinical Score
Description: as for outcome 9
Time Frame: Baseline, Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Score on a scale
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | -1.9 (1.28) | -1.6 (1.22) | -1.8 (1.30)
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | -2.9 (1.27) | -2.8 (1.47) | -2.6 (1.31)
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | -3.2 (1.36) | -3.2 (1.25) | -3.1 (1.25)
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | -3.3 (1.38) | -3.4 (1.06) | -3.3 (1.23)

11. Secondary Outcome: Number of Participants With Modified Clinical Resolution
Description: Modified clinical resolution was defined as a global clinical score of 0 or 1. Global clinical score was defined as the sum of bulbar conjunctival injection and ocular conjunctival discharge scores. Global clinical score was defined as the sum of bulbar conjunctival injection and ocular conjunctival discharge scores. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale.
Time Frame: Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Participants
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | 100 | 28 | 93
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | 166 | 48 | 143
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 189 | 59 | 175
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | 182 | 59 | 173

12. Secondary Outcome: Number of Participants With Expanded Clinical Resolution
Description: Expanded clinical resolution was defined as a global clinical score of 0, 1, or 2 with neither injection nor discharge having a score of 2. Global clinical score was defined as the sum of bulbar conjunctival injection and ocular conjunctival discharge scores. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale.
Time Frame: Day 3, 5, 8 and 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 226 | 76 | 227
Participants
  Day 3: number analyzed (Participants) | 215 | 76 | 218
  Day 3 | 155 | 46 | 154
  Day 5: number analyzed (Participants) | 206 | 65 | 209
  Day 5 | 185 | 54 | 171
  Day 8: number analyzed (Participants) | 205 | 65 | 206
  Day 8 | 193 | 63 | 192
  Day 12: number analyzed (Participants) | 195 | 62 | 187
  Day 12 | 185 | 61 | 181

13. Secondary Outcome: Time to Clinical Resolution
Description: Clinical resolution was defined as absence (score of 0) of bulbar conjunctival injection and ocular conjunctival discharge in the study eye. Bulbar conjunctival injection was assessed based on 0 (Normal conjunctival vascular pattern) - 4 (Markedly prominent, intense diffuse hyperemia) scale which used pictures from VBR scale. Ocular conjunctival discharge was assessed based on 0 (No evidence of discharge in conjunctiva) - 3 (Abundant quantity of mucopurulent or purulent discharge) scale. Time to clinical resolution defined as the date on which a participant first reached clinical resolution minus the date of first dose of investigational product, plus 1.
Time Frame: Baseline to Day 12
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Days | 5 [5.0 to 8.0] | 6 [5.0 to 8.0] | 8 [5.0 to 8.0]

14. Secondary Outcome: Number of Participants Who Used Rescue Medication
Description: Rescue treatment with a licensed antibiotic according to the local standard of care was provided to participants if, in the judgment of the investigator, there was no clinical improvement or worsening of their condition to an extent that it would be in the best interest of the participant treated with an alternate therapy for safety reasons.
Time Frame: Baseline to Day 12
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 223 | 76 | 227
Participants | 2 | 3 | 4

15. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. Any AE that occured after the first dose of investigational product instillation was considered a TEAE.
Time Frame: From start of study drug administration up to 14 days
Population: Safety population included all participants who received at least one dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
Number analyzed (Participants) | 323 | 108 | 321
Participants | 106 | 43 | 61

ADVERSE EVENTS:
Time Frame: From start of study drug administration up to 14 days.
Description: One participant was randomized in error and therefore captured in the ITT population, but not in the Safety Population.
Arm/Group | SHP640 | PVP-I 0.6% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/323 | 0/108 | 0/321
Serious Adverse Events (participants affected / at risk) | 0/323 | 0/108 | 0/321
Other Adverse Events (participants affected / at risk) | 67/323 | 26/108 | 7/321
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP640 (N=323) | PVP-I 0.6% (N=108) | Placebo (N=321)
Instillation site pain (General disorders) | 67 (68) | 26 (26) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (6):
  • Study Protocol: Protocol (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/Prot_000.pdf
  • Study Protocol: Amendment 1 (2016-11-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/Prot_001.pdf
  • Study Protocol: Amendment 2 (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/Prot_002.pdf
  • Study Protocol: Amendment 3 (2017-12-13): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/Prot_003.pdf
  • Study Protocol: Amendment 4 (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/Prot_004.pdf
  • Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/24/NCT03004924/SAP_005.pdf